CLINICAL TRIAL: NCT02167594
Title: 18F-AV-1451 Injection for Brain Imaging of Tau in Subjects With Progressive Supranuclear Palsy (PSP), Subjects With Corticobasal Degeneration (CBD) and Healthy Volunteers
Brief Title: Tau Imaging in Subjects With Progressive Supranuclear Palsy, Corticobasal Degeneration and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A09
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Progressive Supranuclear Palsy; Corticobasal Degeneration
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PSP Subjects (Experimental): Amyloid negative subjects with PSP receiving a flortaucipir PET scan at baseline and at 9 months.
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan
- CBD subjects (Experimental): Amyloid negative subjects with CBD receiving a flortaucipir PET scan at baseline and at 9 months.
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan
- Healthy volunteers (Experimental): Healthy volunteers receiving a flortaucipir PET scan at baseline.
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan

INTERVENTIONS:
Drug: Flortaucipir F18 — IV injection, 370 megabecquerel (MBq) (10 mCi)
  Other Names: [F18]T807; 18F-AV-1451; LY3191748; Tauvid
Procedure: Brain PET scan — positron emission tomography (PET) scan of the brain 75-105 minutes post-injection

SUMMARY:
This study will evaluate flortaucipir for brain imaging of tau in subjects with progressive supranuclear palsy (PSP), corticobasal degeneration (CBD) and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Cognitively Healthy Volunteers

* Mini-mental state examination (MMSE) ≥ 28
* No history of cognitive decline or parkinsonian motor disorder

CBD and PSP subjects

* Able to walk 10 steps with minimal assistance
* MMSE ≥ 14 and ≤ 30
* Subject has a reliable study partner who agrees to accompany subject to visits and spends at least 5 hours per week with the subject

PSP subjects only

* Meet National Institute of Neurological Disorders and Stroke - Society for Progressive Supranuclear Palsy (NINDS-SPSP) probable or possible PSP criteria as modified for the Neuroprotection and Natural History Parkinson Plus Syndromes (NNIPPS) clinical trial

CBD subjects only

* Meets 2013 consensus criteria for possible or probable corticobasal degeneration, corticobasal syndrome (CBS) subtype

Exclusion Criteria:

All subjects

* Have evidence of structural abnormalities such as vascular disease, large strokes or severe white matter disease or other mass lesion on screening MRI
* Claustrophobia
* Current clinically significant cardiovascular disease or clinically significant abnormalities on screening electrocardiogram (e.g. corrected QT interval >450 msec)
* Have a history of risk factors for Torsades de Pointes (e.g. heart failure, hypokalemia, family history of long QT syndrome)
* Have a current clinically significant infectious disease, endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer
* Females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception
* Have received or participated in a trial with investigational medications in the past 30 days
* Have had a non-study related radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session
* Have a history of neuroleptic use for a prolonged period of time or within the past 6 months

PSP and CBD subjects

* Have evidence of amyloid deposition
* Meet National Institute on Aging-Alzheimer's Association criteria for probable Alzheimer's Disease
* Have any other neurological condition other than CBS or PSP that could account for cognitive or motor deficits
* Serum or plasma progranulin level less than one standard deviation below the normal subject mean for the laboratory performing the assay
* Have a high-risk family history suggestive of tar DNA binding protein (TDP)-43 pathology or known mutations

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Avid Radiopharmaceuticals, Inc.
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSD Movement Disorder Clinic, La Jolla, California
  - UCSF Neurosciences Clinical Research Unit, San Francisco, California
  - Molecular Neuroimaging, New Haven, Connecticut
  - Perelman School of Medicine, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited between Aug 2014 and Jul 2016.
Groups:
- PSP Subjects: Amyloid negative subjects with Progressive Supranuclear Palsy (PSP) receiving a flortaucipir PET scan
- CBD Subjects: Amyloid negative subjects with Corticobasal Degeneration (CBD) receiving a flortaucipir PET scan
- Healthy Volunteers: Healthy volunteers receiving a flortaucipir PET scan
Period: Overall Study
Arm/Group | PSP Subjects | CBD Subjects | Healthy Volunteers
Started | 20 | 6 | 3
Completed (Completed = 9 month flortaucipir PET scan acquired) | 18 | 5 | 3
Not Completed | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- PSP Subjects: Amyloid negative subjects with PSP receiving a flortaucipir PET scan at baseline and at 9 months.
  Flortaucipir F18 PET scan: IV injection, 370 MBq (10 mCi)
- CBD Subjects: Amyloid negative subjects with CBD receiving a flortaucipir PET scan at baseline and at 9 months.
  Flortaucipir F18 PET scan: IV injection, 370 MBq (10 mCi)
- Healthy Volunteers: Healthy volunteers receiving a flortaucipir PET scan at baseline.
  Flortaucipir F18 PET scan: IV injection, 370 MBq (10 mCi)
- Total: Total of all reporting groups
Arm/Group | PSP Subjects | CBD Subjects | Healthy Volunteers | Total
Number analyzed (Participants) | 20 | 6 | 3 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (5.88) | 72.2 (7.41) | 68.7 (10.41) | 69.8 (6.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 0 | 10
  Male | 14 | 2 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 19 | 6 | 3 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 18 | 6 | 3 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 6 | 3 | 29
Mini Mental Status Exam (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Mini-mental status exam (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment.
  units on a scale | 26.5 (3.12) | 26.3 (4.32) | 29.3 (0.58) | 26.7 (3.28)

OUTCOME MEASURES:

1. Primary Outcome: Flortaucipir Imaging in PSP, CBD and Healthy Volunteers
Description: A PSP/CBD (PSP = progressive supranuclear palsy; CBD = corticobasal degeneration) targeted composite Standardized Uptake Value ratio (SUVr) was calculated as the voxel-weighted average from the regional SUVr values of the left, right, and total globus pallidus and the dentate nuclei of the cerebellum for both the baseline and 9 month PET scans. Additionally, a global cortical Alzheimer's Disease (AD)-targeted cortical SUVr was calculated. For SUVr, a value of 1 signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain.
Time Frame: baseline and 9 month scans
Population: Healthy volunteers did not receive 9 month follow-up scans. 9 month data presented only for those subjects who completed both a baseline and 9 month scan.
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Groups:
- All Subjects: All subjects combined
Arm/Group | PSP Subjects | CBD Subjects | Healthy Volunteers | All Subjects
Number analyzed (Participants) | 20 | 6 | 3 | 29
standardized uptake value ratio (SUVr)
  Right Dentate Baseline | 1.17 (0.12) | 1.12 (0.04) | 1.03 (0.12) | 1.15 (0.12)
  Right Dentate 9 months: number analyzed (Participants) | 18 | 5 | 0 | 23
  Right Dentate 9 months | 1.17 (0.11) | 1.11 (0.05) |  | 1.15 (0.10)
  Left Dentate Baseline | 1.16 (0.10) | 1.09 (0.04) | 1.08 (0.07) | 1.14 (0.09)
  Left Dentate 9 months: number analyzed (Participants) | 18 | 5 | 0 | 23
  Left Dentate 9 months | 1.13 (0.11) | 1.08 (0.05) |  | 1.12 (0.10)
  Right Globus Pallidus Baseline | 1.60 (0.15) | 1.40 (0.20) | 1.29 (0.06) | 1.53 (0.19)
  Right Globus Pallidus 9 Months: number analyzed (Participants) | 18 | 5 | 0 | 23
  Right Globus Pallidus 9 Months | 1.58 (0.13) | 1.47 (0.19) |  | 1.55 (0.15)
  Left Globus Pallidus Baseline | 1.62 (0.15) | 1.56 (0.32) | 1.30 (0.07) | 1.58 (0.21)
  Left Globus Pallidus 9 Months: number analyzed (Participants) | 18 | 5 | 0 | 23
  Left Globus Pallidus 9 Months | 1.62 (0.15) | 1.62 (0.40) |  | 1.62 (0.21)
  Global PSP/CBD Summary Baseline | 1.38 (0.10) | 1.29 (0.11) | 1.17 (0.03) | 1.34 (0.12)
  Global PSP/CBD Summary 9 Months: number analyzed (Participants) | 18 | 5 | 0 | 29
  Global PSP/CBD Summary 9 Months | 1.37 (0.09) | 1.32 (0.13) |  | 1.36 (0.10)
  AD Cortical Baseline | 0.99 (0.03) | 0.99 (0.06) | 1.02 (0.02) | 0.99 (0.04)
  AD Cortical 9 Months: number analyzed (Participants) | 18 | 5 | 0 | 23
  AD Cortical 9 Months | 0.99 (0.03) | 1.00 (0.05) |  | 0.99 (0.04)

ADVERSE EVENTS:
Time Frame: End of study for AE reporting was 48 hours after flortaucipir administration at each imaging visit.
Description: Adverse Events were defined as occurring or worsening after injection of dose, within 48 hours post injection, at an imaging visit. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to flortaucipir.
Arm/Group | PSP Subjects | CBD Subjects | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 2/20 | 1/6 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PSP Subjects (N=20) | CBD Subjects (N=6) | Healthy Volunteers (N=3)
bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less